CLINICAL TRIAL: NCT00348231
Title: Jikei Optimal Insulin Therapy in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jikei University School of Medicine (Other)
Collaborators: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-195(4220)
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-09-01 (Estimated); Status verified 2006-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus, biphasic insulin analogue
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Drug: dual-action insulin analog

SUMMARY:
The purpose of this study is to compare whether there is the difference in the effect of insulin therapy by the number of times of insulin injection.

DETAILED DESCRIPTION:
The current insulin therapy is divided into the conventional insulin therapy (1~2 injections per day) and the intensive insulin therapy (3~4 injections per day). The kinetics of exogenous insulin in the intensive insulin therapy imitate the kinetics of insulin secretion in a healthy person. A previous large clinical study (e.g. DCCT, Kumamoto study, etc.) suggested that intensive insulin therapy prevented microangiopathy and macroangiopathy, and inhibited progression of them, however many patients chose conventional insulin therapy because many hoped that they injected insulin as few as possible. The patients thought that their life styles were disturbed by many times of insulin injection.

The current dual-acting insulin made from insulin as part modified by protamine is able to suppress postprandial hyperglycemia. The new insulin may possibly have the kinetics of insulin in the patient who uses insulin as the intensive insulin therapy. Moreover, the patients will receive the insulin therapy easily if the times of insulin injection are fewer. It may lead to perform the more effective insulin therapy to search for the optimal insulin therapy in induction in type 2 diabetes.

comparison:HbA1c, glycated albumin, IMT, lipid profile,body weight, daily profile of blood glucose,between the conventional insulin therapy and the intensive insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes
* secondary failure of SU drug
* whose age is to 80 from 20 years old

Exclusion Criteria:

* who has the complication
* who has a allergy of insulin
* who is pregnant

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-11; Study Completion 2006-08

PRIMARY OUTCOMES:
HbA1c
daily profile of blood glucose

SECONDARY OUTCOMES:
IMT
QOL

CONTACTS AND LOCATIONS:
Overall Officials: Yumi Miyashita, MD, Principal Investigator — The Jikei University School of Medicine
Locations (1):
- The Jikei university school of medicine division of diabetes and endoclinology dept. of internal medicine, Tokyo, Tokyo, Japan

REFERENCES:
- [Derived] Miyashita Y, Nishimura R, Nemoto M, Matsudaira T, Kurata H, Yokota T, Yokota K, Tojo K, Utsunomiya K, Tajima N. Prospective randomized study for optimal insulin therapy in type 2 diabetic patients with secondary failure. Cardiovasc Diabetol. 2008 May 29;7:16. doi: 10.1186/1475-2840-7-16. PMID 18507868